CLINICAL TRIAL: NCT05020574
Title: Microbiome and Association With Implant Infections: Investigating the Impact of Antibiotics on the Gut and Breast Microbiomes Post-mastectomy With Implant-based Breast Reconstruction
Brief Title: Microbiome and Association With Implant Infections
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: The Plastic Surgery Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 217510; NCI-2021-08985 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2021-08-20; First posted 2021-08-25 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Breast Cancer Female; Genetic Predisposition to Disease
Keywords: Post-Surgical Antibiotics; Breast Implant Infections; Breast Microbiome; Breast Reconstruction; Mastectomy
MeSH Terms: conditions — Breast Neoplasms; Genetic Predisposition to Disease | interventions — Cephalexin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort A: Standard antibiotics (Experimental): Receive standard pre-incision antibiotics and 24-hour perioperative antibiotics - Prescribed standard postoperative antibiotics to take for at least 7 days post-operatively
  Interventions: Drug: Cephalexin
- Cohort B: No antibiotics (No Intervention): Receive standard pre-incision antibiotics and 24-hour perioperative antibiotics - No antibiotics post-operatively, unless patient develops clinical evidence of infection

INTERVENTIONS:
Drug: Cephalexin — Given orally (PO)
  Other Names: Keflex
  Arms: Cohort A: Standard antibiotics

SUMMARY:
The most common tissue expander-related infections are from Staphylococcus and Pseudomonas species. In addition, from breast tissue microbiome studies, Staphylococcus and Pseudomonas show variable abundance across samples. The investigator hypothesizes that participants undergoing mastectomy with high initial abundance of Staphylococcus and/or Pseudomonas are more likely to develop subsequent tissue expander-related infections from these respective organisms.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility of breast microbiome sampling using the study techniques

SECONDARY OBJECTIVES:

I. To define the differences in the gut and breast microbiomes between participants undergoing mastectomy with implant-based reconstruction who develop post-operative implant infection and those who do not.

II. To determine the effects of post-operative antibiotics on the gut and breast microbiomes after mastectomy with implant-based reconstruction.

OUTLINE: Participants are randomized to 1 of 2 cohorts.

COHORT A: Participants receive postoperative antibiotics to take for at least 7 days post-operatively.

COHORT B: Participants receive no antibiotics post-operatively in the absence of clinical evidence of infection.

Participants are followed up for 90 days.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed breast malignancy OR genetic predisposition to breast cancer.
2. Age >= 18 years
3. Scheduled to undergo mastectomy with the immediate placement of tissue expanders or implant placement
4. Ability to understand a written informed consent document, and the willingness to sign it
5. At least 4 weeks post-completion of chemotherapy or radiation therapy.

Exclusion Criteria:

1. Any significant medical condition or laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
2. Pregnant or breastfeeding
3. Patients who have taken antibiotics within 90 days of the consent date
4. Patients who have taken probiotics within 90 days of the consent date
5. Patients who have a documented or reported allergic reaction to the outlined antibiotics to be used in this study
6. Male patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of tissue samples obtained successfully over time | 90 days
  The feasibility of success in obtaining samples from breast tissue will be measured as a binary outcome (successful or not successful) over time (intra-operatively, week 1, week 2, week 3, and week 4). The investigators will assess and document success in obtaining a tissue sample immediately at the time of sampling of each participant.
Proportion of aspirate samples obtained successfully overall | 90 days
  The feasibility of success in obtaining samples from the tissue expander aspiration ports will be measured as a binary outcome (successful or not successful) over time (intra-operatively, week 1, week 2, week 3, and week 4). The investigators will assess and document success in obtaining a aspirate sample immediately at the time of sampling of each participant.
Proportion of tissue samples successfully producing microbiome data | 90 days
  Feasibility based off of the success rates in producing microbiome data from tissue samples in each patient will be measured as a binary outcome (successful or not successful) and will be reported.
Proportion of aspirate samples successfully producing microbiome data | 90 days
  Feasibility based off of the success rates in producing microbiome data from tissue samples in each patient will be measured as a binary outcome (successful or not successful) and will be reported.
Proportion of any samples successfully producing microbiome data | 90 days
  Feasibility based off of the success rates in producing microbiome data from tissue or aspirate samples in each patient will be measured as a binary outcome (successful or not successful) and will be reported.
Correlation of the change in breast microbiome over time with total duration of antibiotics (Cohort A only) | 90 days
  The investigators will analyze the microbiomes between groups, between microbiome environments (gut v. breast, inter-individual). The correlate of change in breast microbiome over time will be compared to the total duration of antibiotics for Cohort A only. The measure of association ranges from +1 to -1, with a value of zero equal to no association.

SECONDARY OUTCOMES:
Proportion of participants with post-operative infection | 90 days
  Safety will be assessed by clinically assessing for signs of post-operative infection in each patient at each clinic visit. A post-operative infection is defined by clinical assessment of findings of surgical site erythema, tenderness, edema, and/or purulent drainage +/- fever. Proportion of participants with clinically diagnosed infection will be reported for each group and final diagnosis for analyses will be binary; a participant will either have a post-operative infection in the 90 day post-operative period or not have a post-operative infection in the 90 day post-operative period.
Shannon Diversity Index Score for species of microbiome | 90 days
  Alpha diversity will be evaluated for species richness by number of operational taxonomic units and for evenness using the Shannon Index. The Shannon diversity index (H) is an index that is commonly used to characterize species diversity in a community and accounts for both abundance and evenness of the species present. The proportion of species (i) relative to the total number of species (pi) is calculated, and then multiplied by the natural logarithm of this proportion (lnpi). The resulting product is summed across species, and multiplied by -1. Shannon's equitability (EH) can be calculated by dividing H by Hmax (here Hmax = lnS). Equitability assumes a value between 0 and 1 with 1 being complete evenness and the overall index score is represented by a percentage of the species.
Number of overall identified microbes | 90 days
  The investigators will evaluate microbial composition by grouping identified microbes into operational taxonomic units at the species, genera and phyla levels and will compare the relative abundances of these microbes between groups at the species, gene

CONTACTS AND LOCATIONS:
Overall Officials: Merisa Piper, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No